CLINICAL TRIAL: NCT05955365
Title: Monotherapy With a P2Y12 Inhibitor Followed by a Direct-acting Oral Anticoagulant in Patients With ATRial fIbrillation Undergoing suprafleX Cruz Coronary Stent Implantation
Brief Title: Monotherapy With P2Y12 Inhibitors in Patients With Atrial fIbrillation Undergoing Supraflex Stent Implantation
Acronym: MATRIX-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Sahajanand Medical Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MATRIX-2
Record Dates: First submitted 2023-06-28; First posted 2023-07-21 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Percutaneous Coronary Intervention (PCI); Atrial Fibrillation (AF); Oral Anticoagulation; P2Y12 Inhibitor
MeSH Terms: conditions — Atrial Fibrillation | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monotherapy strategy (Experimental): Patients randomized to the monotherapy treatment arm receive any of the commercially available oral P2Y12 inhibitors (clopidogrel, prasugrel oder ticagrelor) and immediately discontinue aspirin and DOAC (or will not re-start DOAC after PCI if treatment was temporarily stopped before). After 1 month, the P2Y12 inhibitor will be stopped and treatment with a commercially available DOAC (at investigator's discretion and dosed according to the instructions for use in patients with atrial fibrillation) will be initiated for the duration of 11 months. After completion of the 12-month study regimen (study visit), the patient will receive antithrombotic therapy according to routine care.
  Interventions: Drug: P2Y12 inhibitor; Drug: DOAC
- Standard of care strategy (Active Comparator): Patients randomized to the standard of care, receive DOAC for at least 12 months. In addition, aspirin is administered for up to 1 month after PCI at investigator's discretion and one of the available P2Y12 inhibitors (clopidogrel, prasugrel oder ticagrelor at investigator's discretion) is administered for a minimum of 6 months and up to 12 months after PCI. After completion of the 12-month control arm regimen (study visit), the patients will be treated according to routine care.
  Interventions: Drug: P2Y12 inhibitor; Drug: Aspirin; Drug: DOAC

INTERVENTIONS:
Drug: P2Y12 inhibitor — The choice of P2Y12 inhibitor is left at investigator's discretion.
Drug: Aspirin — Aspirin is administered for up to 1 month after PCI at investigator's discretion
  Arms: Standard of care strategy
Drug: DOAC — The choice of DOAC is left at investigator's discretion.

SUMMARY:
Patients with atrial fibrillation undergoing percutaneous coronary intervention with stent implantation require treatment with different antithrombotic drugs. Oral anticoagulants are prescribed to reduce the risk of stroke associated with atrial fibrillation. Antiplatelet substances are prescribed after stent implantation to reduce the risk of adverse cardiac events such as myocardial infarction or stent thrombosis. Treatment with antithrombotic medications can cause bleeding complications, particularly when these substances are combined.

The currently recommended standard strategy consists of treatment with 3 antithrombotic medications for at least 1 week up to one month, followed by treatment with two of these medications for up to 6-12 months after stent implantation. Thereafter, patients usually receive long-term treatment with only one drug, an anticoagulant.

In the monotherapy group of this study, the investigators will investigate a strategy where only one antithrombotic drug will be used at a time. During the first month after stent implantation, the investigators will prescribe an antiplatelet medication, followed by an oral anticoagulant as monotherapy. This strategy might be associated with fewer bleeding complications, while protecting adequately against thrombotic events.

In this study the investigators would like to investigate whether treatment with a single antithrombotic drug ("monotherapy strategy") is associated with benefits compared to the currently recommended combination therapy of antithrombotic medications ("standard-of-care strategy").

DETAILED DESCRIPTION:
Background:

The optimal antithrombotic treatment following percutaneous coronary intervention (PCI) in patients with atrial fibrillation (AF) requiring long-term oral anticoagulation remains a matter of debate. In particular, the appropriate intensity and duration of antithrombotic strategies to prevent ischemic events, while mitigating the risk of bleeding complications in this high bleeding risk population during the early peri-procedural period (within 30 days) and thereafter (from 30 days to 1 year) following drug-eluting stent implantation remains unclear.

Aim:

The investigators aim to assess the safety and efficacy of a P2Y12 inhibitor monotherapy regimen for 1 month followed by DOAC monotherapy long-term versus current standard of care consisting of triple antithrombotic therapy for up to one month (aspirin, P2Y12 inhibitor and DOAC) followed by dual antithrombotic therapy (P2Y12 inhibitor and DOAC) for 6 to 12 months and DOAC monotherapy thereafter, in AF patients undergoing PCI indicated for treatment with a DOAC after sirolimus-eluting Supraflex Cruz stent implantation and followed for a period of 12 months.

Methodology:

This investigator-initiated, multi-center, randomized, open-label, blinded evaluation, international clinical trial in 3010 AF patients with indication for long-term oral anticoagulation who have undergone successful PCI with Supraflex Cruz sirolimus-eluting biodegradable polymer cobalt chromium stent implantation. The study will be conducted at approximately 150 sites across Europe and Brazil. Patients will be randomized to the antithrombotic monotherapy (experimental antithrombotic strategy) or the standard of care strategy (control group) in a 1:1 ratio. Randomization is stratified by site, acute coronary syndrome (ACS) within the previous 6 months and CHA2DS2-VASc score ≥4. Patients randomized to the antithrombotic monotherapy treatment receive any of the commercially available oral P2Y12 inhibitors (clopidogrel, ticagrelor, prasugrel) and immediately discontinue aspirin and DOAC. After 1 month, the P2Y12 inhibitor will be stopped and treatment with a commercially available DOAC will be initiated for the duration of 11 months. Patients randomized to the standard of care strategy will initiate triple therapy for up to 1 month followed by dual anti-thrombotic therapy (consisting of P2Y12 inhibitor for a minimum of 6 and up to 12 months plus DOAC for at least 12 months).

Potential significance:

This is the first study investigation the impact of a short course of P2Y12 inhibitor monotherapy up to 1 month, while omitting clopidogrel non-responders, and temporarily omitting OAC, after stent implantation followed by OAC monotherapy in AF patients undergoing PCI. This sequential monotherapy treatment strategy has solid rational and carries potential to balance bleeding against cardiac and cerebral ischemic risks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Atrial fibrillation or flutter with an indication for oral anticoagulation using direct-acting oral anticoagulants (DOACs) for ≥12 months
* Successful percutaneous coronary intervention in at least 1 lesion within the previous 7 days with no remaining lesions intended for treatment.
* Free from major adverse events post qualifying PCI, including new onset chest pain suspected to be of ischemic origin, acute or subacute stent thrombosis, new-onset neurological signs or symptoms.
* Written informed consent

Exclusion Criteria:

* Planned staged percutaneous intervention procedure (Patients can be enrolled after complete coronary revascularization with no remaining lesions intended for treatment. Patients who have or develop indication to percutaneous valve intervention can undergo treatment more than 30 days after qualifying PCI.)
* Cardioversion for treatment of atrial fibrillation within 1 month prior to inclusion or planned cardioversion
* AF ablation procedure within 2 months prior to inclusion or planned AF ablation procedure
* Prior mechanical valvular prosthesis implantation
* Deep vein thrombosis/pulmonary embolism, at least moderately severe mitral stenosis or other clinical conditions than atrial fibrillation requiring long-term oral anticoagulation
* Stroke within 1 month prior to randomization
* Hemodynamic instability (persistent systolic blood pressure below 90 mmHg, continuous infusions of catecholamines, clinical signs of hypoperfusion and/or use of percutaneous left ventricular assist devices)
* Uncontrolled severe hypertension with a systolic blood pressure (BP) ≥180 mmHg and/or diastolic BP ≥120 mmHg
* Severe renal impairment with estimated creatinine clearance (CrCL) <15 mL/min or on dialysis
* Moderate or severe hepatic impairment (Child-Pugh Class B or C) or any hepatic disease associated with coagulopathy
* Any hypersensitivity or contraindications for direct oral anticoagulation or dual antiplatelet therapy with aspirin and a P2Y12 inhibitor
* Any of the following abnormal local laboratory results prior to randomization: platelet count <50 x109/L or hemoglobin <8 g/dL
* Known pregnancy or breast-feeding patients
* Life expectancy <1 year due to other severe non-cardiac disease
* Planned surgery including coronary artery bypass grafting within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3010 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of participants with a major adverse cardiac or cerebral events (MACCE), defined as the composite of death from any cause, myocardial infarction, stroke or non-central nervous system (non-CNS) systemic embolism | 12 months
The number of participants with a major or clinically relevant non-major bleeding (MCB), defined according to the International Society of Thrombosis and Haemostasis (ISTH) criteria | 12 months

SECONDARY OUTCOMES:
The incidence of MACCE or MCB | 12 months
  MACCE, defined as the composite of death from any cause, myocardial infarction, stroke or non-CNS systemic embolism and MCB, defined according to the ISTH criteria
The incidence of MACCE or MCB | 15 months
  MACCE, defined as the composite of death from any cause, myocardial infarction, stroke or non-CNS systemic embolism and MCB, defined according to the ISTH criteria
The number of participants with a composite of death from cardiovascular causes, myocardial infarction or stroke | 12 months
The number of participants with a composite of death from cardiovascular causes, myocardial infarction or stroke | 15 months
The number of participants with a composite of death from cardiovascular causes, myocardial infarction, stroke or non-CNS systemic embolism | 12 months
The number of participants with a composite of death from cardiovascular causes, myocardial infarction, stroke or non-CNS systemic embolism | 15 months
The number of participants died from cardiovascular or non-cardiovascular causes | 12 months
The number of participants died from cardiovascular or non-cardiovascular causes | 15 months
The number of participants with a composite of stroke and non-CNS systemic embolism | 12 months
The number of participants with a composite of stroke and non-CNS systemic embolism | 15 months
The number of participants with any stroke (including ischemic, hemorrhagic and unknown types) | 12 months
The number of participants with any stroke (including ischemic, hemorrhagic and unknown types) | 15 months
The number of participants with an ischaemic stroke | 12 months
The number of participants with an ischaemic stroke | 15 months
The number of participants with a hemorrhagic stroke | 12 months
The number of participants with a hemorrhagic stroke | 15 months
The number of participants with a transient ischemic attack | 12 months
The number of participants with a transient ischemic attack | 15 months
The number of participants with a composite of definite or probable stent thrombosis | 12 months
The number of participants with a composite of definite or probable stent thrombosis | 15 months
The number of participants with a definite stent thrombosis | 12 months
The number of participants with a definite stent thrombosis | 15 months
The number of participants with a hospitalization | 12 months
The number of participants with a hospitalization | 15 months
The number of participants with a composite of death or hospitalization | 12 months
The number of participants with a composite of death or hospitalization | 15 months
The number of participants with any target lesion revascularization | 12 months
The number of participants with any target lesion revascularization | 15 months
The number of participants with any target vessel revascularization | 12 months
The number of participants with any target vessel revascularization | 15 months
The number of participants with any revascularization | 12 months
The number of participants with any revascularization | 15 months
The number of all bleeding events, also adjudicated according to Bleeding Academic Research Consortium, Thrombolysis in Myocardial Infarction or Global Use of Strategies to Open Occluded Coronary Arteries scales | 12 months
  The BARC is scaled from 0 to 5, with higher scores indicating worse outcomes, the TIMI from minor to major to fatal bleeding, and the GUSTO from mild to moderate to severe or life-threatening.
The number of all bleeding events, also adjudicated according to Bleeding Academic Research Consortium, Thrombolysis in Myocardial Infarction or Global Use of Strategies to Open Occluded Coronary Arteries scales | 15 months
  The BARC is scaled from 0 to 5, with higher scores indicating worse outcomes, the TIMI from minor to major to fatal bleeding, and the GUSTO from mild to moderate to severe or life-threatening.
Transfusion rates both in patients with and/or without clinically detected overt bleeding | 12 months
Transfusion rates both in patients with and/or without clinically detected overt bleeding | 15 months
The number of participants with a major adverse cardiac or cerebral events (MACCE), defined as the composite of death from any cause, myocardial infarction, stroke or non-central nervous system (non-CNS) systemic embolism | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, Prof, Principal Investigator — Bern University Hospital, Department of Cardiology; Marco Valgimigli, Prof, Principal Investigator — Cardiocentro Ticino Institute
Locations (15):
- Hartcentrum Hasselt, Hasselt, Belgium
- CHU Nîmes, Nîmes, France
- Germany (2):
  - Universitätsklinikum Frankfurt/Main, Frankfurt am Main
  - Klinikum Friedrichshafen, Friedrichshafen
- Italy (2):
  - Ospedale Ferrarotto, Catania, Catania CT
  - IRCCS Humanitas, Milan, Rozzano
- UMC public, Amsterdam, Netherlands
- Uniwersytet Medyczny im. Karola Marcinkowskiego w Poznaniu, Poznan, Poland
- Hospital Universitario Marques de Valdecilla, Santander, Spain
- Switzerland (5):
  - Cardiocentro Ticino Institute, Lugano, Canton Ticino
  - Universitätsspital Basel, Basel
  - Inselspital, Bern University Hospital, Department of Cardiology, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - University Hospital Zürich, Zurich
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No